CLINICAL TRIAL: NCT01410357
Title: Improving Outcomes for Individuals With Serious Mental Illness and Diabetes
Acronym: TTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Martha Sajatovic, MD, Professor of Psychiatry, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01MH085665 (NIH); R01MH085665 (NIH)
Record Dates: First submitted 2011-07-29; First posted 2011-08-05 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus; Bipolar Disorder; Depression; Psychotic Disorders; Schizophrenia
Keywords: serious mental illness; diabetes
MeSH Terms: conditions — Diabetes Mellitus; Bipolar Disorder; Depression; Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Targeted Training in Illness Management (TTIM) (Experimental): Participants in this arm will receive the TTIM intervention as well as receiving regular treatment for their DM and SMI from their normal medical and mental health care providers.
  Interventions: Behavioral: Targeted Training in Illness Management (TTIM)
- Treatment As Usual (TAU) (No Intervention): Participants in this arm will continue to receive Treatment as Usual from their usual medical and mental health care providers. They will not receive any intervention.

INTERVENTIONS:
Behavioral: Targeted Training in Illness Management (TTIM) — This intervention blends psychoeducation, problem identification/goal-setting, behavioral modeling and reinforcement via use of Peer Educators, and health care linkage, has been adapted to the primary care setting and targeted for SMI-DM participants. Generalizability is enhanced with relatively brief in-person participation requirements and by utilizing professional staff typically found in primary care. TTIM will stress information sharing that is accessible to participants, and through a collaborative process, foster motivation for SMI-DM self-management.
  Arms: Targeted Training in Illness Management (TTIM)

SUMMARY:
This project tests a model for improving illness self-management among persons who have both serious mental illness and diabetes and will be performed within a primary care setting at a safety net hospital system. The information gained from the randomized trial will be supplemented with reports from participants about their experiences of trying to improve illness self-management. Improvements in self-management should result in a reduction of psychiatric symptoms and improvements in functioning and physical health.

DETAILED DESCRIPTION:
This project will test a novel intervention, Targeted Training in Illness Management (TTIM), intended to improve both serious mental illness (SMI) and diabetes mellitus (DM) self-management in 100 individuals with SMI-DM vs. 100 individuals with SMI-DM receiving treatment as usual (TAU). The intervention will be conducted in a safety-net health system primary care setting and will be conducted as a randomized controlled trial (RCT). The primary effects of TTIM will be assessed with respect to SMI symptoms, Functional Status/Role Impairment, General Health Status, and DM outcomes. Secondary outcomes include adherence to psychotropic and DM medication, and engagement in healthy behaviors.

This assessment will include quantitative assessment of facilitators/barriers targeted by the proposed intervention as well as a supplemental qualitative assessment. The qualitative assessments will include input from patients and interventionists. Specific aims for the qualitative analysis are to validate findings from the RCT, expand understanding of "key active ingredients" of TTIM, and provide information to inform future studies on individuals with SMI and related medical conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Have Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder or major depression
2. Have DM based upon either previous diagnosis or laboratory values
3. Be ≥ 18 years of age
4. Be able to communicate in English
5. Be able to provide written, informed consent to participation.

Exclusion Criteria:

1. Actively suicidal/homicidal
2. Unable to be rated on study rating scales
3. Demented
4. Pregnant
5. Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — Case Western Reserve University; Neal V Dawson, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make deidentified data available to other qualified investigators in the research community. Data will remain under control of the PIs of the research study at CWRU. Copies of electronic data files accompanied by data documentation (metadata) will be shared.
  Qualified investigators may contact the PIs for information on how to request data. Investigators will be required (at minimum) to provide 1) the names and qualifications of all individuals who will have any access to primary data files; 2) a research proposal detailing how the data will be used; 3) a statement that the investigators will a) not further share the primary data with third parties, b) protect the privacy of subjects, c) provide a means to protect the confidentiality of the data; and 4) a data transfer/use agreement with CWRU. Only data necessary to meet the goals of the investigators' research proposal will be provided to limit the risk of identifying individual research subjects.

REFERENCES:
- [Derived] Sajatovic M, Howland M, Gunzler D, Kanuch SW, Cassidy KA, McCormick R, Bauer MS, Scheidemantel T, Thomas C, Blixen C, Dawson NV. Race analysis in an African American sample with serious mental illness and comorbid diabetes. Psychiatr Rehabil J. 2018 Sep;41(3):246-252. doi: 10.1037/prj0000314. PMID 30160510
- [Derived] Aftab A, Bhat C, Gunzler D, Cassidy K, Thomas C, McCormick R, Dawson NV, Sajatovic M. Associations among comorbid anxiety, psychiatric symptomatology, and diabetic control in a population with serious mental illness and diabetes: Findings from an interventional randomized controlled trial. Int J Psychiatry Med. 2018 May;53(3):126-140. doi: 10.1177/0091217417749795. Epub 2017 Dec 27. PMID 29280685

RESULTS

PARTICIPANT FLOW:
Groups:
- Targeted Training in Illness Management (TTIM): Participants in this arm received the TTIM intervention as well as regular treatment for their DM (diabetes mellitus) and SMI (serious mental illness) from their normal medical and mental health care providers.
  Targeted Training in Illness Management (TTIM): This intervention blended psychoeducation, problem identification/goal-setting, behavioral modeling and reinforcement via use of Peer Educators, and health care linkage, and was adapted to the primary care setting and targeted SMI-DM participants. Generalizability was enhanced with relatively brief in-person participation requirements and professional staff typically found in primary care were utilized. TTIM stressed information sharing that is accessible to participants, and through a collaborative process, fostered motivation for SMI-DM self-management.
- Treatment As Usual (TAU): Participants in this arm received Treatment as Usual from their usual medical and mental health care providers. They did not receive any intervention.
Period: Overall Study
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Started | 100 | 100
Completed | 74 | 76
Not Completed | 26 | 24
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 23 | 21

BASELINE CHARACTERISTICS:
Groups:
- Targeted Training in Illness Management (TTIM): Participants in this arm received the TTIM intervention as well as regular treatment for their DM and SMI from their normal medical and mental health care providers.
  Targeted Training in Illness Management (TTIM): This intervention blended psychoeducation, problem identification/goal-setting, behavioral modeling and reinforcement via use of Peer Educators, and health care linkage, and was adapted to the primary care setting and targeted SMI-DM participants. Generalizability was enhanced with relatively brief in-person participation requirements and professional staff typically found in primary care were utilized. TTIM stressed information sharing that is accessible to participants, and through a collaborative process, fostered motivation for SMI-DM self-management.
- Total: Total of all reporting groups
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU) | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (9.7) | 52.6 (9.7) | 52.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 65 | 128
  Male | 37 | 35 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 38 | 36 | 74
  African-American | 52 | 55 | 107
  Other | 10 | 9 | 19
  Hispanic | 10 | 7 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100 | 100 | 200
Education [Mean (Standard Deviation); unit: years] | 12.7 (2.5) | 12.5 (2.9) | 12.6 (2.7)
Health Insurance Type [Count of Participants; unit: Participants]
  Private | 5 | 2 | 7
  Medicare | 35 | 34 | 69
  Medicaid | 48 | 47 | 95
  Other/None | 12 | 17 | 29
Mini-International Neuropsychiatric Interview (MINI) [Count of Participants; unit: Participants]
  Schizophrenia | 29 | 20 | 49
  Bipolar Disorder | 22 | 34 | 56
  Major Depressive Disorder | 49 | 46 | 95
Serious Mental Illness duration [Mean (Standard Deviation); unit: years] | 19.1 (12.9) | 17.8 (12.4) | 18.5 (12.6)
Diabetes mellitus duration [Mean (Standard Deviation); unit: years] | 9.8 (7.5) | 10.3 (8.1) | 10.1 (7.8)
AHA-defined hypertension [Count of Participants; unit: Participants] | 45 | 42 | 87
On second generation antipsychotic medication [Count of Participants; unit: Participants] | 40 | 33 | 73
Insulin user [Count of Participants; unit: Participants] | 43 | 45 | 88
Charlson Index [Mean (Standard Deviation); unit: scores on a scale] — The self-reported Charlson Index evaluates medical comorbidity. Possible scores range from 0 to 9, with higher scores indicating higher comorbidity. There are no subscales for this measure, just a total score that is summed.
  scores on a scale | 2.4 (1.7) | 2.1 (1.5) | 2.2 (1.6)
Basic Health Literacy Screen [Mean (Standard Deviation); unit: scores on a scale] — The Basic Health Literacy Scale is comprised of three items on a 5-point response scale, ranging from 1-5. After reverse-scoring the item addressing confidence with forms (item #2), responses to the three items are summed. Total scores range between 3 and 15, with higher scores indicating higher subjective health literacy.
  scores on a scale | 12.5 (3.0) | 12.4 (3.3) | 12.5 (3.2)
Clinical Global Impression [Mean (Standard Deviation); unit: scores on a scale] — The Clinical Global Impression (CGI) is a broad measure of global psychopathology that evaluates illness severity on a 1 to 7 point continuum. Possible scores range from 0 to 7, with higher scores indicating greater psychopathology.
  scores on a scale | 4.3 (1.0) | 4.3 (0.9) | 4.3 (0.9)
Montgomery Asberg Depression Rating Scale [Mean (Standard Deviation); unit: scores on a scale] — The MADRS is a 10-item depression severity scale widely utilized in studies with patients with serious mental illness. Possible scores range from 0 to 60 with higher scores indicating worse depression.
  scores on a scale | 23.1 (9.4) | 25.0 (8.8) | 24.1 (9.1)
Brief Psychiatry Rating Scale [Mean (Standard Deviation); unit: scores on a scale] — The BPRS measures psychotic and non-psychotic symptoms in serious mental illness. Possible total scores range from 7 to 126, with higher scores indicating greater symptom severity. For this study, the BPRS with 18 items was used. Each symptom measured ranges from 1-7, and all 18 items/symptoms are summed to create the total score. Only the BPRS total score was utilized in the analyses.
  scores on a scale | 38.7 (9.8) | 41.3 (8.9) | 40.0 (9.3)
Global Assessment of Functioning [Mean (Standard Deviation); unit: scores on a scale] — The GAF is a 100-point single-item scale that measures global functioning. Possible scores range from 1 to 100, with higher scores indicating better functioning.
  scores on a scale | 51.8 (11.0) | 51.4 (11.9) | 51.6 (11.5)
Sheehan Disability Scale [Mean (Standard Deviation); unit: scores on a scale] — The SDS measures role impairment in three domains (work/school; family life/home; social life). Possible total scores range from 0 to 30, with higher scores indicating greater disability. Only the total score was reported in our analyses, and is denoted here. The total score is calculated by summing the three domain scores, each which range from 0-10.
  scores on a scale | 18.0 (5.8) | 17.8 (6.5) | 17.9 (6.2)
Short-form 36 (general health status) [Mean (Standard Deviation); unit: scores on a scale] — The Short Form 36 Health Survey (SF-36) is a self-report of general health divided into a physical component summary (PCS) and mental component summary (MCS). Norm-based scores are placed on the same metric with a mean of 50 and standard deviation of 10. Scores above 50 reflect higher functional status than the average population and scores below 50 reflect lower than average function. Both the physical and mental are separate subscales with their own scoring as determined by the process above.
  scores on a scale
    Physical | 39.4 (10.1) | 39.8 (10.9) | 39.6 (10.5)
    Mental | 37.2 (10.6) | 35.6 (12.1) | 36.4 (11.4)
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: mmol/mol] | 8.2 (2.0) | 8.0 (2.4) | 8.2 (2.3)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 135.0 (20.7) | 134.5 (21.7) | 134.8 (21.2)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 35.4 (8.0) | 36.6 (9.4) | 36.0 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Brief Psychiatric Rating Scale (BPRS) at 60 Weeks
Description: The BPRS measures psychotic and non-psychotic symptoms in serious mental illness. Possible total scores range from 7 to 126, with higher scores indicating greater symptom severity. For this study, the BPRS with 18 items was used. Each symptom measured ranges from 1-7, and all 18 items/symptoms are summed to create the total score. Only the BPRS total score was utilized in the analyses.
Time Frame: 60 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 74 | 76
scores on a scale | 32.04 (9.0) | 35.89 (8.7)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM); Test type: Superiority; p = .785, Mixed Models Analysis — Bonferroni corrections were conducted to adjust for multiple comparisons

2. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS) at 60 Weeks
Description: The MADRS is a 10-item depression severity scale widely utilized in studies with patients with serious mental illness. Possible scores range from 0 to 60 with higher scores indicating worse depression.
Time Frame: 60 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 74 | 76
scores on a scale | 15.92 (10.0) | 18.55 (8.8)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .016, Mixed Models Analysis; A Bonferroni correction was conducted to adjust for multiple comparisons

3. Primary Outcome: Clinical Global Impression (CGI) at 60 Weeks
Description: The Clinical Global Impression (CGI) is a broad measure of global psychopathology that evaluates illness severity on a 1 to 7 point continuum. Possible scores range from 0 to 7, with higher scores indicating greater psychopathology.
Time Frame: 60 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 74 | 76
scores on a scale | 3.24 (1.1) | 4.03 (1.1)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p < 0.001, Mixed Models Analysis; A Bonferroni correction was conducted to adjust for multiple comparisons

4. Primary Outcome: Global Assessment of Functioning (GAF) at 60 Weeks
Description: The GAF is a 100-point single-item scale that measures global functioning. Possible scores range from 1 to 100, with higher scores indicating better functioning.
Time Frame: 60 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 74 | 76
scores on a scale | 61.05 (13.1) | 53.29 (13.3)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .003, Mixed Models Analysis; A Bonferroni correction was conducted to adjust for multiple comparisons

5. Primary Outcome: Sheehan Disability Scale (SDS) at 60 Weeks
Description: The SDS measures role impairment in three domains (work/school; family life/home; social life). Possible total scores range from 0 to 30, with higher scores indicating greater disability. Only the total score was reported in our analyses, and is denoted here. The total score is calculated by summing the three domain scores, each which range from 0-10.
Time Frame: 60 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 74 | 76
scores on a scale | 15.0 (7.4) | 16.47 (7.1)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .086, Mixed Models Analysis

6. Primary Outcome: SF-36 (Short-form) Health Survey at 60 Weeks; Mental Health Component
Description: The Short Form 36 Health Survey (SF-36) is a self-report of general health divided into a physical component summary (PCS) and mental component summary (MCS). Norm-based scores are placed on the same metric with a mean of 50 and standard deviation of 10. Scores above 50 reflect higher functional status than the average population and scores below 50 reflect lower than average function.
Time Frame: 60 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 74 | 76
scores on a scale | 42.05 (11.1) | 39.58 (11.4)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .872, Mixed Models Analysis; A Bonferroni correction was conducted to adjust for multiple comparisons

7. Primary Outcome: Glycosylated Hemoglobin (HbA1c) at 60 Weeks
Time Frame: 60 weeks
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 74 | 76
mmol/mol | 7.69 (1.9) | 7.77 (2.0)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .662, Mixed Models Analysis

8. Primary Outcome: Systolic Blood Pressure at 60 Weeks
Time Frame: 60 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 74 | 76
mmHg | 134.12 (20.7) | 132.71 (23.8)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .633, Mixed Models Analysis

9. Primary Outcome: Body Mass Index (BMI) at 60 Weeks
Time Frame: 60 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 74 | 76
kg/m^2 | 36.46 (8.6) | 37.07 (9.8)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .175, Mixed Models Analysis; A Bonferroni correction was conducted to adjust for multiple comparisons

10. Primary Outcome: SF-36 Health Survey at 60 Weeks; Physical Health Component
Description: as for outcome 6
Time Frame: 60 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 74 | 76
scores on a scale | 39.65 (11.1) | 40.81 (9.3)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .680, Mixed Models Analysis; A Bonferroni correction was conducted to adjust for multiple comparisons

11. Secondary Outcome: Tablets Routine Questionnaire (TRQ) at 60 Weeks
Description: The self-reported Tablets Routine Questionnaire (TRQ) measures change in treatment adherence. The TRQ determines proportion of prescribed medication missed, and ranges from 0 (no medication missed/100% adherent) to 100 (no medication taken/0% adherent). The TRQ format captured an exact proportion (%) of days with a missed medication dose for each oral maintenance psychotropic medication and then an average combined TRQ was calculated for all orally-prescribed medications.
Time Frame: 60 weeks
Measure: Mean (Standard Deviation); unit: percentage of days adherent
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 74 | 76
percentage of days adherent | 17.09 (30.19) | 18.65 (30.10)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .407, Mixed Models Analysis

12. Secondary Outcome: Self-rated Diabetes Self-Care Activities (SDSCA) Questionnaire at 60 Weeks
Description: The SDSCA measure is a brief self-report questionnaire of diabetes self-management that includes items assessing the following aspects of the diabetes regimen: general diet, specific diet, exercise, blood-glucose testing, foot care, and smoking. It is comprised of 10 questions, to which each have a 5 point scale with anchors 1= never through 5= always. The items are summed to a total score, which ranges from 10-50.
Time Frame: 60 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 74 | 76
scores on a scale | 47.69 (20.40) | 48.28 (18.73)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .870, Mixed Models Analysis

13. Secondary Outcome: Comparison of AUDIT (Alcohol Use Disorders Identification Test) Score Between TTIM and TAU (Treatment as Usual) at 60 Weeks
Description: The AUDIT scale (Alcohol Use Disorders Identification Test) has 10 questions, with scores on each question ranging from 0 to 4 (0= never, 1= less than monthly, 2= monthly, 3= weekly 4= daily/almost daily). Questions 9 and 10 only have three anchors: 0, 2, and 4. The scores are summed to get total. Therefore, the range of possible scores are 0-40, with higher scores indicating indicating a greater likelihood of hazardous and harmful drinking. However, such scores may also reflect greater severity of alcohol problems and dependence, as well as a greater need for more intensive treatment.
Time Frame: 60 weeks
Population: While 74 participants completed the TTIM arm and 76 completed TAU, there was some missing data for this scale, resulting in 69 TTIM and 73 TAU.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 69 | 73
Scores on a scale | 1.93 (5.23) | 1.16 (2.57)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .707, Mixed Models Analysis

14. Secondary Outcome: Comparison of ISMI (Internalized Stigma of Mental Illness -Alienation) Between TTIM and TAU at 60 Weeks
Description: The ISMI (Internalized Stigma of Mental Illness) has 29 questions, broken into 5 subscales. This subscale, Alienation, has 6 Likert-scale items. Each question is rated as 1= strongly disagree, 2= disagree, 3= neutral, 4= agree, 5= strongly agree. Total scores on the Alienation subscale range from 6-30, with higher scores reflecting higher levels of reported internalized stigma of mental illness.
Time Frame: 60 weeks
Population: While 74 participants completed the TTIM arm and 76 completed TAU, there was some missing data for this scale, resulting in 70 TTIM and 74 TAU.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 70 | 74
scores on a scale | 15.41 (4.91) | 15.55 (6.07)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .838, Mixed Models Analysis

15. Secondary Outcome: Comparison of ISMI (Stereotype Endorsement) Score Between TTIM and TAU at 60 Weeks
Description: The ISMI (Internalized Stigma of Mental Illness) has 29 questions, broken into 5 subscales. This subscale, Stereotype Endorsement, has 7 Likert-scale items. Each question is rated as 1= strongly disagree, 2= disagree, 3= agree, 4= strongly agree. Total scores on the Stereotype Endorsement subscale range from 7-28, with higher scores reflecting higher levels of reported internalized stigma of mental illness.
Time Frame: 60 weeks
Population: While 74 participants completed the TTIM arm and 76 completed TAU, there was some missing data for this scale, resulting in 69 TTIM and 74 TAU.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 69 | 74
scores on a scale | 13.80 (3.27) | 13.92 (3.86)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .853, Mixed Models Analysis

16. Secondary Outcome: Comparison of ISMI (Discrimination Experience) Between TTIM and TAU at 60 Weeks
Description: The ISMI (Internalized Stigma of Mental Illness) has 29 questions, broken into 5 subscales. This subscale, Discrimination Experience, has 5 Likert-scale items. Each question is rated as 1= strongly disagree, 2= disagree, 3= neutral, 4= agree, 5= strongly agree. Total scores on the Discrimination Experience subscale range from 5-25, with higher scores reflecting higher levels of reported internalized stigma of mental illness.
Time Frame: 60 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 70 | 74
scores on a scale | 12.63 (4.47) | 12.31 (4.82)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .853, Mixed Models Analysis

17. Secondary Outcome: Comparison of ISMI (Social Withdrawal) Score Between TTIM and TAU at 60 Weeks
Description: The ISMI (Internalized Stigma of Mental Illness) has 29 questions, broken into 5 subscales. This subscale, Social Withdrawal, has 6 Likert-scale items. Each question is rated as 1= strongly disagree, 2= disagree, 3= neutral, 4= agree, 5= strongly agree. Total scores on the Social Withdrawal subscale range from 6-30, with higher scores reflecting higher levels of reported internalized stigma of mental illness.
Time Frame: 60 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 70 | 74
scores on a scale | 14.50 (4.71) | 13.85 (4.98)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .510, Mixed Models Analysis

18. Secondary Outcome: Comparison of ISMI (Stigma Resistance) Score Between TTIM and TAU at 60 Weeks
Description: The ISMI (Internalized Stigma of Mental Illness) has 29 questions, broken into 5 subscales. This subscale, Stigma Resistance, has 5 Likert-scale items. Each question is rated as 0= strongly disagree, 1= disagree, 2= neutral, 3= agree, 4= strongly agree. These scores are all reverse coded. Total scores on the Stigma Resistance subscale range from 0-20, with higher scores reflecting higher levels of reported internalized stigma of mental illness.
Time Frame: 60 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 70 | 74
scores on a scale | 5.84 (2.86) | 6.47 (3.34)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .573, Mixed Models Analysis

19. Other Pre Specified Outcome: Comparison of Utilization (Phys Ed) Score Between TTIM and TAU at 60 Weeks
Description: The Utilization of Physical Education score looks at how many times a participant used these resources. Analyses include a simple mean and SD.
Time Frame: 60 weeks
Population: While 74 participants completed the TTIM arm and 76 completed TAU, there was some missing data for this scale, resulting in 74 TTIM and 75 TAU.
Measure: Mean (Standard Deviation); unit: times utilized
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 74 | 75
times utilized | .85 (2.43) | .65 (.94)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .758, Mixed Models Analysis

20. Other Pre Specified Outcome: Comparison of Utilization (Mental Ed) Score Between TTIM and TAU at 60 Weeks
Description: The Utilization of Mental Education score looks at how many times a participant used these resources. Analyses include a simple mean and SD.
Time Frame: 60 weeks
Population: While 76 completed TAU, there was some missing data for this scale, resulting in 74 TAU.
Measure: Mean (Standard Deviation); unit: times utilized
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 74 | 74
times utilized | .03 (.16) | .00 (.00)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .156, Mixed Models Analysis

21. Other Pre Specified Outcome: Comparison of Utilization (Mental Hospital) Score Between TTIM and TAU at 60 Weeks
Description: The Utilization of Mental Hospital score looks at how many times a participant used these resources. Analyses include a simple mean and SD.
Time Frame: 60 weeks
Population: While 74 participants completed the TTIM arm and 76 completed TAU, there was some missing data for this scale, resulting in 73 TTIM and 74 TAU.
Measure: Mean (Standard Deviation); unit: time utilized
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 73 | 74
time utilized | .03 (.16) | .00 (.00)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .156, Mixed Models Analysis

22. Other Pre Specified Outcome: Comparison of Diabetes Knowledge Score Between TTIM and TAU at 60 Weeks
Description: The diabetes knowledge score has 23 questions which assess how much knowledge one has about diabetes. They are in multiple choice format, with 4 choices, and only one is correct. The total amount correct is added up, and then calculated into a percentage of answers correct.
Time Frame: 60 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 73 | 74
percent correct | 74.57 (16.59) | 63.02 (20.58)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p < .001, Mixed Models Analysis

23. Other Pre Specified Outcome: Comparison of MSPSS (Multidimensional Scale of Perceived Social Support) Score Between TTIM and TAU at 60 Weeks
Description: The Multidimensional Scale of Perceived Social Support is a 12 question Likert scale, with each item ranging from 1-5. Total scores range from 12-60, with higher scores indicating more perceived social support.
Time Frame: 60 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 73 | 74
scores on a scale | 44.11 (8.45) | 43.69 (9.54)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .878, Mixed Models Analysis

24. Other Pre Specified Outcome: Comparison of PDSMS (Perceived Diabetes Self Management Scale)Score Between TTIM and TAU at 60 Weeks
Description: The Perceived Diabetes Self-Management Scale is an 8-item Likert scale, with each question ranging from 1-5. Items 1, 2, 6, and 7 are reverse coded. Total summed scores range from 8-40, with higher scores indicating higher perceived self-management competence in regards to diabetes.
Time Frame: 60 weeks
Population: While 74 participants completed the TTIM arm and 76 completed TAU, there was some missing data for this scale, resulting in 67 TTIM and 72 TAU.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 67 | 72
scores on a scale | 29.66 (4.74) | 26.76 (7.48)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .014, Mixed Models Analysis

25. Other Pre Specified Outcome: Comparison of PMHSMS (Perceived Mental Health Self-Management Scale) Score Between TTIM and TAU at 60 Weeks
Description: The Perceived Mental Health Self-Management Scale is an 8-item Likert scale, with each question ranging from 1-5. Total summed scores range from 8-40, with higher scores indicating higher perceived self-management competence in regards to mental health.
Time Frame: 60 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
Number analyzed (Participants) | 70 | 74
scores on a scale | 28.43 (5.76) | 26.86 (7.21)
Statistical Analysis 1: Comparison: Targeted Training in Illness Management (TTIM) vs Treatment As Usual (TAU); Test type: Superiority; p = .227, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Targeted Training in Illness Management (TTIM) | Treatment As Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 2/100 | 1/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No